CLINICAL TRIAL: NCT01081353
Title: An Open Label 4-Way Crossover Pharmacokinetic Trial of New Formula Aspirin Versus Effervescent Aspirin in Healthy Adult Subjects
Brief Title: Pharmacokinetic Study Comparing Aspirin and Effervescent Aspirin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14961
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Pharmacokinetics
Keywords: Aspirin; Acetylsalicylic Acid
MeSH Terms: interventions — Aspirin; Glutaredoxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin BAY1019036)
- Arm 2 (Active Comparator)
  Interventions: Drug: Alka Seltzer Extra Strength
- Arm 3 (Active Comparator)
  Interventions: Drug: Aspirin Migraine
- Arm 4 (Active Comparator)
  Interventions: Drug: Aspirin Aspro

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin BAY1019036) — One tablet of new formula Aspirin under fasting conditions
  Arms: Arm 1
Drug: Alka Seltzer Extra Strength — One effervescent tablet under fasting conditions
  Arms: Arm 2
Drug: Aspirin Migraine — One effervescent tablet under fasting conditions
  Arms: Arm 3
Drug: Aspirin Aspro — One effervescent tablet under fasting conditions
  Arms: Arm 4

SUMMARY:
To determine the bioequivalence of new formula of aspirin relative to the established commercial effervescent aspirin when taken orally by healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 to 55 years of age inclusive with a Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs)
* Results of screening and clinical laboratory tests are within normal range or considered not clinically significant by the Principal Investigator or Sponsor
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, Depo-Provera, or a double barrier and have a negative pregnancy test at Screening and Day 0 for each Dosing Period. Female subjects of non-childbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy
* Be willing to participate in all scheduled visits, treatment plan, laboratory tests and other trial procedures according to the clinical protocol

Exclusion Criteria:

* History of hypersensitivity to aspirin (ASA), Nonsteroidal Antiinflammatory Drugs (NSAIDs), acetaminophen and similar pharmacological agents or components of the products
* Eighteen to twenty year olds with a viral infection, with or without fever, at the time of dosing - Syndromes of asthma, rhinitis or nasal polyps
* Females who are pregnant or lactating
* Have taken ASA, ASA-containing products, acetaminophen or any other NSAID (Over the counter (OTC) or prescription) 7 days prior to dosing or during the treatment period, other than trial treatment
* Smokers or currently consuming any type of tobacco product(s) including any smoking cessation nicotine-containing product (e.g., nicotine patch, nicotine gum)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Bioavailability of new formulation aspirin versus marketed effervescent tablets (500mg aspirin) | 24 hours

SECONDARY OUTCOMES:
Adverse event collection | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hackensack, New Jersey, United States